CLINICAL TRIAL: NCT02183272
Title: Ketamine as an Adjunctive Treatment of Acute Suicidal Ideation in the Emergency Setting.
Brief Title: Emergency Ketamine Treatment of Suicidal Ideation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Cheryl McCullumsmith, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ketamine IIT
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Depression; Suicidal Ideation; Suicidal Impulses
Keywords: Depression; Suicidal Ideation; Ketamine; Emergency Department
MeSH Terms: conditions — Depression; Suicidal Ideation; Emergencies | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Ketamine (Active Comparator): 0.2 mg / kg dose of intranasal ketamine for treatment of suicidality will be given in two separate doses on the day of admission to the hospital.
  Interventions: Drug: Intranasal Ketamine
- Intranasal Saline Placebo (Placebo Comparator): 0.2 mg / kg dose saline intranasal will be given in two separate doses on the day of hospital admission.
  Interventions: Drug: Intranasal Saline Placebo

INTERVENTIONS:
Drug: Intranasal Ketamine — Ketamine in liquid form to be distributed nasally by a board-certified physician while the subject is already in the hospital for suicidal ideation.
  Other Names: ketamine
  Arms: Intranasal Ketamine
Drug: Intranasal Saline Placebo — Intranasal Saline to be distributed by a board-certified physician while the patient is already hospitalized for suicidal ideation.
  Other Names: saline
  Arms: Intranasal Saline Placebo

SUMMARY:
The objective of the current program of research will be to test whether intranasal ketamine treatment is more effective than placebo in reducing suicidal ideation in suicidal patients presenting for acute treatment in emergency department settings. Secondary objectives will test the effect of genotypic differences in the mu opioid receptor on efficacy of ketamine and the correlation of speech patterns and facial movement patterns with subjective reductions in suicidal ideation after ketamine treatment.

DETAILED DESCRIPTION:
The objective of the current program of research will be to test whether intranasal ketamine treatment is more effective than placebo in reducing suicidal ideation in suicidal patients presenting for acute treatment in emergency department settings. Secondary objectives will test the effect of genotypic differences in the mu opioid receptor on efficacy of ketamine and the correlation of speech patterns and facial movement patterns with subjective reductions in suicidal ideation after ketamine treatment

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Ages 18-65
3. All races and ethnicities
4. Willing and able to provide informed consent
5. A cutoff score of >3 on the Beck Scale for Suicidal Ideation
6. >2 on the Columbia Scale for Suicide Severity Rating

Exclusion Criteria:

1. Pregnancy or lactation; women of reproductive potential must have a negative urine pregnancy test
2. Post-partum state (within 2 months of delivery)
3. Homicide risk as determined by clinical interview
4. Any of the following Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnoses:

   1. Any current primary psychotic disorder
   2. Acute intoxication or withdrawal from alcohol or any other substance of abuse, as determined by clinical interview and urine drug screen except opioids
   3. use of any hallucinogen (except cannabis), in the last month
   4. Any dissociative disorder
   5. Pervasive developmental disorder
   6. Cognitive disorder
   7. Cluster A personality disorder
   8. Anorexia nervosa.
5. Treatment with any medication known to affect the N-methyl-D-aspartate (NMDA) receptor system (e.g., lamotrigine, acamprosate, memantine, riluzole, or lithium)
6. Any known hypersensitivity or serious adverse effect with ketamine
7. Any clinically-significant medication or condition that would preclude the use of ketamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-11 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Ketamine effect on Suicidal Ideation and Depression. | 4 weeks
  To assess the acute efficacy and durability of effect over a 4 week time period of single dose of 0.2 mg/kg intranasal ketamine treatment on suicidal ideation and depression in individuals with acute suicidal ideation as measured by the Beck Scale for Suicidal Ideation (BSS) and the Montgomery-Asberg Depression Rating Scale (MADRS)as compared to placebo.

SECONDARY OUTCOMES:
Assessment of Role of Mu Opioid Receptor | 4 weeks
  To assess the role of specific mu opioid receptor genetic variants in prediction of response to ketamine to alleviate suicidal ideation.

OTHER OUTCOMES:
Assessment of Changes of Biological Markers | 4 weeks
  To assess the changes in biological markers of suicide risk such as linguistic patterns, voice and facial movements after ketamine treatment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl McCullumsmith, MD PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Domany Y, McCullumsmith CB. Single, Fixed-Dose Intranasal Ketamine for Alleviation of Acute Suicidal Ideation. An Emergency Department, Trans-Diagnostic Approach: A Randomized, Double-Blind, Placebo-Controlled, Proof-of-Concept Trial. Arch Suicide Res. 2022 Jul-Sep;26(3):1250-1265. doi: 10.1080/13811118.2021.1878078. Epub 2021 Feb 14. PMID 33583341